CLINICAL TRIAL: NCT00796861
Title: Phase II Pilot Efficacy Trial of Sunitinib for Refractory Malignant Ascites
Brief Title: Trial of Sunitinib for Refractory Malignant Ascites
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Phycisican decided to terminate study due to slow patient accrual.
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Leah Cream, Assistant Professor of Medicine, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSHCI25224
Record Dates: First submitted 2008-11-21; First posted 2008-11-24 (Estimated); Results first posted 2017-12-20 (Actual); Last update posted 2017-12-20 (Actual); Status verified 2017-12

CONDITIONS: Ascites
Keywords: malignant ascites
MeSH Terms: conditions — Ascites | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm (Experimental): Sunitinib (50mg PO daily x 4 wks + 2 wks rest x 3 cycles if able to tolerate tx
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Sunitinib — Patients will be given Sunitinib 50 mg orally daily for four weeks, followed by a two week holiday. For patients tolerating treatment, three cycles of treatment will be given (18 weeks total).
  Other Names: Sunitinib malte

SUMMARY:
The study is to see whether treatment with Sunitinib decreases the accumulation of ascites in patients with refractory malignant ascites.

DETAILED DESCRIPTION:
This is a single arm, non-randomized, phase II pilot study in patients who have stopped cytotoxic and biologic therapy for their neoplasms and are suffering from malignant ascites that requires drainage for comfort. The study will employ a Simon 2-stage optimal design. Initially up to 17 patients would be enrolled. If there are no responses among the first 12 patients, the study would be terminated. Otherwise the trial would be expanded by 23 to a total of 37 patients. If there are 3 or fewer responses by the end of the trial, then no further investigation would be warranted.

ELIGIBILITY:
Inclusion Criteria:

* Solid tumor malignancy and failure of at least one biologic or cytotoxic regimen, or the inability to receive standard treatment due to performance status (PS>2).
* Ascites based on paracentesis or CT scan within one month prior to enrollment
* Life expectancy > 3 months
* Indwelling paracentesis catheters are permitted, paracentesis is permitted at the investigators discretion
* Negative urine pregnancy test for females
* All subjects must agree to use birth control
* All subjects must abstain from eating grapefruit and grapefruit juice. They must tell their physicians about any changes in their medication including over-the-counter and herbal supplements.

Exclusion Criteria:

* History of congestive heart failure
* Creatinine > 2.0
* Pregnant or nursing
* ALT > 2.5 times the upper limit of normal
* Blood pressure > 160/90 (antihypertensives permitted)
* Gastrointestinal or intra-abdominal hemorrhage within the last 6 months
* History of QTc > 450 milliseconds
* Brain metastasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2007-05; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leah Cream, MD, Principal Investigator — Penn State University
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Not enough valuable data

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Arm
Started | 4
Completed | 0
Not Completed | 4
Not completed — Withdrawal by Subject | 2
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate Where a Response is Considered to be 3 cm or More Decrease in Abdominal Girth.
Description: A response will be considered to be 3 cm or more decrease in abdominal girth, or decreased frequency of paracentesis (compared to pre-enrollment). Toxicity monitoring would be the same as that is the expanded access Sutent trial.
Time Frame: An average of every 6 weeks
Population: No analyses were performed as none of the subjects made it through a full cycle.
Arm/Group | Single Arm
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: 1 subject withdrew consent before beginning treatment; only 3 subjects participated in treatment.
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 3/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=3)
Weakness (General disorders) | 1 (1)
Nausea (General disorders) | 2 (4)
Fatigue (General disorders) | 1 (1)
Vomiting (General disorders) | 2 (3)
Decreased appetite (General disorders) | 1 (1)
Erythematous macular erruption (Skin and subcutaneous tissue disorders) | 1 (1)
Insomnia (General disorders) | 1 (1)
Tremors (General disorders) | 1 (1)
Feeling cold (General disorders) | 1 (1)
Stenotrophomas (3+) lesion right thigh (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulcers (Skin and subcutaneous tissue disorders) | 1 (1)
Increased creatinine level (Renal and urinary disorders) | 1 (1)
Increased aspartate aminotransferase (AST) level (Hepatobiliary disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
UTI (General disorders) | 1 (1)
Labial exoriation (Skin and subcutaneous tissue disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Anorexia (General disorders) | 1 (1)
Hyponatremia (General disorders) | 1 (1)
Hyperkalemia (General disorders) | 2 (2)
Hypocalcemia (General disorders) | 2 (2)
Decreased Albumin level (General disorders) | 1 (1)
Hypoglycemia (General disorders) | 2 (2)
Increased Hemoglobin count (General disorders) | 1 (1)
Decreased white blood cell count (General disorders) | 1 (1)
Decreased platelet count (General disorders) | 1 (1)
Ulcer (Skin and subcutaneous tissue disorders) | 1 (4)
Fissures (Skin and subcutaneous tissue disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less